CLINICAL TRIAL: NCT06983535
Title: Induction of Labor (IOL) Using Cervical Double-balloon (Cook Catheter) in Outpatient Versus Inpatient Setting (COOK Study): a Multicentre, Randomised Controlled Trial.
Brief Title: Comparing Outpatient and Inpatient Use of a Cervical Balloon for Starting Labor in Low-Risk Pregnancies.
Acronym: Cook
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusion rate
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: AZ Sint-Lucas Brugge (Other); University Hospital, Antwerp (Other); Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GYN2016.01
Record Dates: First submitted 2025-04-24; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Induction of Labor
Keywords: induction of labor; cervical ripening; balloon catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Inpatient (Active Comparator): Patient in this arm were randomized to stay in the hospital during cervical balloon ripening
  Interventions: Device: cervical balloon catheter
- Outpatient (Active Comparator): Patients in this arm were randomized to ambulant home setting during cervical ripening
  Interventions: Device: cervical balloon catheter

INTERVENTIONS:
Device: cervical balloon catheter — Patients will be randomized to inpatient or outpatient setting while having the cervical ripening balloon catheter

SUMMARY:
Why was this study done? About 20-30% of pregnancies involve labor being started artificially, known as induction. One way to do this is with a balloon catheter placed in the cervix, which helps prepare the body for labor. This mechanical method works just as well as using medication but may be safer for the baby, as it reduces the chances of the womb contracting too much (which can cause stress to the baby). Because it's safe and simple, this method could possibly be done at home instead of in the hospital.

What was the aim of the study? The researchers wanted to compare how safe and effective this balloon method is when used at home (outpatient) versus in the hospital (inpatient). They also wanted to know how satisfied women were with each approach.

How was the study done? The study took place at four hospitals in Belgium between 2017 and 2023. It included women with healthy low risk pregnancies who were scheduled for induction for non-urgent reasons, such as being past their due date, having a large baby, or by personal choice after 38 weeks of pregnancy.

The women were randomly placed into two groups:

Outpatient setting: going home after balloon placement.

Inpatient setting: staying in the hospital after balloon placement<

The main thing researchers measured was whether the baby's heart rate pattern (checked by CTG monitoring) was abnormal after 12 hours. They also looked at how the baby was born (vaginal birth or C-section), how long labor took, whether additional medicine was needed, pain management, and how satisfied the mothers were with the process.

DETAILED DESCRIPTION:
Study Design and Approval

This was a randomised controlled trial - a scientific study designed to compare two groups as fairly as possible. It took place in four hospitals in Belgium:

Ziekenhuis Oost-Limburg (ZOL), Genk

AZ Sint-Lucas, Brugge

Jessa Ziekenhuis, Hasselt

University Hospital Antwerp (UZA), Antwerp

The study ran from May 2017 to November 2023. It was carefully reviewed and approved by the Ethics Committee of ZOL Genk and the review boards of the other hospitals to make sure it followed strict ethical and safety standards.

Who Could Take Part?

Women were eligible to join the study if they:

Were over 18 years old

Were pregnant with just one baby

Had a baby in the head-down (cephalic) position

Had a Bishop Score of 6 or less (indicating the cervix wasn't ready for labor)

Needed their labor to be induced for low-risk reasons, such as:

Being past their due date (post-term)

Suspected large baby (macrosomia)

Personal request to induce labor after 38 weeks of pregnancy

Women were not allowed to join the study if they had any of the following:

Twins or more (multiple pregnancy)

Preterm premature rupture of membranes (water breaking too early)

A baby not growing well (fetal growth restriction)

A condition called placenta accreta spectrum (PAS)

A previous cesarean section

Baby not in head-down position

Gestational diabetes or high blood pressure during pregnancy

Lived more than 60 minutes away from the hospital

Any other health issues (maternal or fetal) or reason that made vaginal birth unsafe

How Were Women Assigned to Groups? Women were told about the study by their doctor in the days leading up to labor induction. On the day of induction, a hospital doctor checked if they met the criteria. If they did, the woman was asked to sign a consent form to take part in the study.

Once enrolled, each woman was randomly assigned to one of two groups:

Inpatient group - stayed in the hospital after balloon insertion

Outpatient group - went home after balloon insertion

The randomisation was done using a computer program, so neither the doctors nor patients could influence which group they were placed into. Because it was obvious who went home and who stayed, this study was not blinded.

The Induction Procedure All four hospitals had experience using mechanical methods to start labor. Before the study began, all staff received a brief training guide to ensure the procedure was done the same way in every hospital.

How the Balloon Was Inserted:

A double-balloon catheter (Cook balloon) was gently inserted into the cervix using a special tool under direct view with a vaginal speculum.

The lower balloon (inside the uterus) was first filled with 20 ml of saline.

The balloon was pulled back so that it rested properly in the cervix.

Then both balloons (one inside the uterus and one in the vagina) were gradually filled with saline up to 80 ml each.

The catheter was taped to the woman's thigh to keep it in place, but no tension or pulling was applied.

After insertion, each woman was monitored for 2 hours using CTG to check the baby's heart rate and any contractions.

If the CTG after balloon insertion was not normal (e.g., slow heartbeat, signs of stress), the woman stayed in the hospital, even if she was in the outpatient group.

Outpatient Group: Going Home If the CTG was normal, women in the outpatient group went home with the balloon still in place and were asked to return to the hospital 12 hours later, unless one of the following happened: their water broke (spontaneous rupture of membranes), they started having strong or painful contractions, the balloon came out or moved, they experienced non-tolerable pain or felt anxious, they simply didn't want to go home.

Before going home, every woman was given clear, written instructions about: when to come back early, what warning signs to look for, how to call the hospital, they also received a follow-up call from the doctor on duty 1-2 hours after leaving, to check how they were doing.

After 12 Hours: Balloon Removal and Next Steps. Twelve hours after the balloon was placed (or sooner, if needed), the balloon was removed. At that time the Bishop Score was checked again to see if the cervix had softened or opened. A new CTG was performed to make sure the baby was doing well.

What happened next depended on how the cervix looked: if the cervix was still not ready (Bishop Score ≤ 6):

→ Labor was continued using prostaglandins (a medication to soften the cervix)

If the cervix was ready (Bishop Score > 6) and effaced (thinned out):

→ Labor was started by breaking the water (amniotomy) and giving oxytocin to strengthen contractions

If the cervix was open but not thinned, doctors often chose oral or vaginal prostaglandins instead of breaking the water.

All clinical details were recorded by trained hospital staff.

Primary Outcome (Main Focus):

The baby's wellbeing as seen on the CTG (heart rate monitor) right after the balloon was inserted and again when it was removed (or sooner if problems occurred).

Secondary Outcomes (Other Important Measures):

1. Maternal Clinical Outcomes:

   How the baby was delivered (normal, assisted with vacuum or forceps, cesarean)

   Pain relief used (e.g., paracetamol, pethidine, epidural)

   Use of labor medications like oxytocin
2. Process Outcomes:

   How long the entire induction process took:

   From hospital admission to discharge

   From balloon placement to delivery

   From balloon removal to delivery
3. Maternal Satisfaction:

   Assessed using a detailed 16-question survey sent by email 1-2 days after delivery

   Topics included overall experience, comfort, timing, and whether they'd choose the same method again
4. Maternal Health Concerns:

Possible complications like:

Uterine hyperstimulation (too many contractions)

Placental abruption (placenta detaching early)

Infections needing antibiotics

Doctors also recorded why some women needed C-sections or assisted births.

ELIGIBILITY:
Inclusion Criteria:

* women >18 years of age with singleton pregnancies, cephalic presentation and a unfavourable cervix requiring priming (Bishop Score ≤ 6) that needed an IOL for low risk indications: post-term, macrosomia, patient's preference (> 38 0/7 weeks of gestational age).

Exclusion Criteria:

* : multiple pregnancies, preterm premature rupture of membranes (pPROM), foetal growth restriction (FGR), placenta-accreta spectrum (PAS), previous C-Section(s), non-cephalic presentation, gestational diabetes, hypertensive disorders of pregnancy, living at >60 minutes from the hospital, any other maternal or foetal morbidity, any other contraindication to vaginal birth.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Fetal wellbeing | 12 hours
  The primary outcome was foetal wellbeing assessed by cardiotocography (CTG) immediately after balloon insertion and balloon removal (12 hours after insertion). The CTG could be normal or not normal. The CTG was reported as not normal in case of a baseline rise, decelerations (even if they were not repeated decelerations) or decreased variability. The second CTG assessment was performed earlier in case of vaginal bleeding, fluid loss, onset of regular painful contractions, balloon expulsion or in any other case judged clinically relevant by the obstetrician

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Pieters, Study Chair — Data Science Institute, Hasselt University, Diepenbeek, Belgium.
Locations (4):
- Belgium (4):
  - University Hospitals Antwerp, Antwerp, Antwerp
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Jessa Ziekenhuis, Hasselt, Limburg
  - AZ Sint Lucas, Bruges, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: Yes
Data regarding the different outcomes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 05/2017-11/2043
Access Criteria: Only the central study team will have access

REFERENCES:
- [Background] Alfirevic Z, Keeney E, Dowswell T, Welton NJ, Medley N, Dias S, Jones LV, Caldwell DM. Methods to induce labour: a systematic review, network meta-analysis and cost-effectiveness analysis. BJOG. 2016 Aug;123(9):1462-70. doi: 10.1111/1471-0528.13981. Epub 2016 Mar 22. PMID 27001034
- See also: European Perinatal Health Report: Core Indicators of the Health and Care of Pregnant Women and Babies in Europe from 2015 to 2019. Euro-Peristat — https://www.europeristat.com/publications/european-perinatal-health-report-2015-2019/